CLINICAL TRIAL: NCT03335722
Title: Investigating Non-invasive Brain Stimulation to Enhance Fluency in People Who Stutter
Acronym: INSTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R52173/RE001_
Record Dates: First submitted 2017-10-26; First posted 2017-11-08 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Stuttering, Developmental
Keywords: stammering; speech motor disorder; electrical current stimulation; metronome-timed speech
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled (sham tDCS), randomised trial, with 20 participants with developmental stuttering recruited for each of the two arms of the trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A researcher from another research group who is not involved in any aspect of the trial will perform the randomisation of participants into the sham and tDCS study arms using a minimisation procedure within "randPack" package in R (Carey and Gentleman, 2016). Allocation concealment will be achieved by assigning a unique 5-digit code per participant (containing no identifying information regarding trial arm). This will be emailed to the researcher. The code is used to deliver stimulation via study mode on the stimulator (http://www.neurocaregroup.com/dc_stimulator_plus.html). The participants and the researchers who will deliver the intervention, assess the outcomes, and analyse the data will be masked to trial arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TDCS and Fluency Intervention (Active Comparator): Participants will receive 1-milliamp (mA) tDCS with the anode (5 x 7 cm) placed over the left frontal cortex and the cathode (5 x 7 cm) placed symmetrically over the right frontal cortex. tDCS will be delivered using a direct current (DC) stimulator in 'study-mode' for 20 minutes a day for five consecutive days. he stimulation will be applied for the first half of a 40-minute speech fluency training paradigm, using metronome-timed speech.
  Interventions: Behavioral: Metronome-timed speech; Device: Active tDCS
- Sham TDCS and Fluency Intervention (Sham Comparator): Participants will receive sham stimulation with the anode and cathode electrodes placed over the left and right frontal cortex as in the active arm. Sham stimulation will be delivered using a DC-stimulator in 'study-mode' for 20 minutes a day for five consecutive days. For sham stimulation, the current is ramped up over 15 seconds, maintained for 15 seconds at 1 mA and ramped down over 15 seconds at the start of stimulation and is then followed by brief (3ms) pulses every 55 seconds for the remainder of the 20-minute stimulation session. he stimulation will be applied for the first half of a 40-minute speech fluency training paradigm, using metronome-timed speech.
  Interventions: Behavioral: Metronome-timed speech; Device: Sham tDCS

INTERVENTIONS:
Behavioral: Metronome-timed speech — Reading, narrative, and conversational speech tasks will be completed on each of the five intervention days. Metronome- timed speech will be practiced during these tasks, at near-normal (comfortable) speech rate for each participant. Each intervention session will be 40 minutes in duration.
Device: Active tDCS — 1-mA tDCS with the anode (5 x 7 cm) placed over the left frontal cortex and the cathode (5 x 7 cm) placed symmetrically over the right frontal cortex. tDCS will be delivered using a direct current (DC) stimulator in 'study-mode' for 20 minutes. The current is ramped up to 1 mA over the first 15 seconds of stimulation and maintained at this level for remainder of the 20-minute stimulation session.
  Arms: Active TDCS and Fluency Intervention
Device: Sham tDCS — Sham stimulation will be delivered using a DC-stimulator in 'study-mode' for 20 minutes. Participants will receive sham stimulation with the anode and cathode electrodes placed over the left and right frontal cortex as in the active arm. For sham stimulation, the current is ramped up over 15 seconds, maintained for 15 seconds at 1 mA and ramped down over 15 seconds at the start of stimulation and is then followed by brief (3ms) pulses every 55 seconds for the remainder of the 20-minute stimulation session.
  Arms: Sham TDCS and Fluency Intervention

SUMMARY:
This study aims to test whether the application of transcranial direct current stimulation (tDCS) concurrent with fluency training results in improvements in speech fluency in adults with developmental stuttering, measured up to three months after the intervention.

DETAILED DESCRIPTION:
Developmental stuttering affects 5% of children and persists to adulthood in about 1%. Changing the way speech is produced in adults who stutter is a particular challenge for speech and language therapy and there is a need for novel interventions. One such intervention involves the application of transcranial direct current stimulation (tDCS) alongside therapies aimed at improving speech fluency. tDCS influences brain activity by modulating neuronal plasticity through the application of weak electrical currents across the brain. Pairing tDCS with speech therapy has potential for producing larger or longer lasting effects and reducing time spent in therapy.

The study will evaluate the potential of tDCS combined with speech fluency training to improve outcomes in people who stutter (PWS). PWS will have this training while receiving tDCS for five days (1 milliampere [mA] for 20 mins per day) in a double-blind randomized controlled trial. Outcomes will be measured in terms of changes to stuttering severity.

An additional research questions is how changes in interactions between sensory and motor brain regions relate to changes in speech fluency in PWS. MRI will be used to measure brain structure and function and the vocal tract during speech production. Transcranial magnetic stimulation (TMS) will assess motor excitability before and after the training.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Diagnosed with developmental stuttering of mild-moderate or greater severity
* Native speaker of English
* Normal or corrected-to-normal vision
* Normal hearing

Exclusion Criteria:

* Speech, language or communication disorder other than developmental stuttering.
* Contraindication to brain stimulation (tDCS or TMS)
* Contraindication to MRI
* History of drug abuse
* History of a neurological or psychiatric illness
* Any previous neurosurgical procedures
* Taking prescription or over-the-counter medication that may affect brain function (for example, anti-depressants)
* Family history of epilepsy (first degree relative)
* Severe claustrophobia (as they may be unable to tolerate scanner)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Stuttering Severity Instrument (SSI-4) Score | 1 week, 6 weeks and 12 weeks after the end of the 5-day intervention
  The Stuttering Severity Instrument (SSI-4) is a standardised measure of stuttering severity comprised of 3 sub-scores (frequency, duration and physical concomitants) which are summed to give a total score. We will use change from baseline in total score (i.e. baseline subtracted) on the Stuttering Severity Instrument version 4 measured post intervention. The maximum total score of the SSI-4 is 56, which corresponds to the highest stuttering severity. Therefore, larger negative change scores represent better outcomes (larger reductions in stuttering severity).

SECONDARY OUTCOMES:
Change in percentage of disfluent syllables produced during conversation | 1 week, 6 weeks and 12 weeks after the end of the 5-day intervention
  Change from baseline (i.e. baseline subtracted) in percentage of disfluent syllables produced during a two-minute conversation sample. Larger negative change scores represent better outcomes (larger reductions in frequency of disfluency).
Change in percentage of disfluent syllables produced during reading | 1 week, 6 weeks and 12 weeks after the end of the 5-day intervention
  Change from baseline (i.e. baseline subtracted) in percentage of disfluent syllables produced during a two-minute reading sample. Larger negative change scores represent better outcomes (larger reductions in frequency of disfluency).
Change in Overall Assessment of the Speaker's Experience of Stuttering (OASES) score | 6 weeks and 12 weeks after the end of the 5-day intervention
  The Overall Assessment of the Speaker's Experience of Stuttering (OASES) is a standardised self-assessment to measure the effect of stuttering on a person's life, comprising of 4 sub-scores (general information about speech, your reactions to stuttering, communication in daily situations, quality of life). The total score (out of a possible 500) is divided by the number of items (out of a possible 100. Note that some items may not apply to all participants). This gives a total impact score between 1 and 5, with 5 representing the highest negative impact on person's life.
  We will use change from baseline in total score (i.e. baseline subtracted) on the OASES total impact score, measured post intervention, as an outcome. Larger negative change scores represent better outcomes (larger reductions in negative impact of stuttering ).

OTHER OUTCOMES:
Change in Premonitory Awareness in Stuttering Scale | 1 week, 6 weeks and 12 weeks after the end of the 5-day intervention
  Change in total score on measure of anticipation of stuttering
Change in Beck Anxiety Inventory | 1 week, 6 weeks and 12 weeks after the end of the 5-day intervention
  Change in total score on the Beck Anxiety Inventory
Change in Subjective rating of stuttering severity | 1 week, 6 weeks and 12 weeks after the end of the 5-day intervention
  Change in self-rating on 9 point scale
Change in Subjective rating of speech naturalness | 1 week, 6 weeks and 12 weeks after the end of the 5-day intervention
  Change in self-rating on 9 point scale
Change in Objective rating of stuttering severity | 1 week, 6 weeks and 12 weeks after the end of the 5-day intervention
  Change in Researcher rating on 9 point scale
Change in Objective rating of speech naturalness | 1 week, 6 weeks and 12 weeks after the end of the 5-day intervention
  Change in Researcher rating on 9 point scale

CONTACTS AND LOCATIONS:
Overall Officials: Kate E Watkins, PhD, Principal Investigator — University of Oxford
Locations (1):
- Department of Experimental Psychology, University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: INSTEP trial website — https://insteptrial.wordpress.com
- See also: Speech and Brain Research Group website — https://www.psy.ox.ac.uk/research/speech-brain-research-group

DOCUMENTS (3):
  • Study Protocol (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT03335722/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT03335722/SAP_003.pdf
  • Informed Consent Form (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT03335722/ICF_002.pdf